CLINICAL TRIAL: NCT00053248
Title: A Phase I/II Study To Determine The Safety, Tolerability, And Anti-Leukemic Effects of Trisenox (Arsenic Trioxide) In Combination With Gleevec (STI571) In Patients With Resistant Chronic Myelogenous Leukemia In Chronic Phase
Brief Title: Arsenic Trioxide and Imatinib Mesylate in Treating Patients With Chronic Myelogenous Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000269319; OHSU-UCLA-0206062; OHSU-HEM-02001-L; OHSU-1096
Record Dates: First submitted 2003-01-27; First posted 2003-01-28 (Estimated); Last update posted 2012-05-28 (Estimated); Status verified 2010-06

CONDITIONS: Leukemia
Keywords: chronic phase chronic myelogenous leukemia; Philadelphia chromosome positive chronic myelogenous leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Arsenic Trioxide; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: arsenic trioxide
Drug: imatinib mesylate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Imatinib mesylate may stop the growth of cancer cells by blocking the enzymes necessary for cancer cell growth. Combining chemotherapy with imatinib mesylate may kill more cancer cells.

PURPOSE: Phase I/II trial to study the effectiveness of combining arsenic trioxide with imatinib mesylate in treating patients who have chronic phase chronic myelogenous leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and tolerability of arsenic trioxide and imatinib mesylate in patients with resistant chronic phase chronic myelogenous leukemia.
* Determine potential dose-limiting toxic effects in patients treated with this regimen.
* Determine the pharmacokinetics of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive oral imatinib mesylate once daily and arsenic trioxide IV over 1-2 hours on days 1-5 of week 1 and then twice weekly. Treatment continues for 1 year in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 18-24 patients (at least 6 patients for phase I and at least 12 patients for phase II) will be accrued for this study .

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Cytogenetically confirmed Philadelphia chromosome-positive (Ph+) chronic myelogenous leukemia, meeting one of the following criteria:

  * Chronic phase

    * Less than 15% blasts in peripheral blood or marrow
    * Less than 30% blasts and promyelocytes in peripheral blood or marrow
    * Less than 20% basophils in blood or marrow
    * Platelet count at least 100,000/mm^3 (unless therapy related)
    * No progressive (increase of at least 10 cm in any 4 of the past 24 weeks) or existing (greater than 10 cm) splenomegaly
  * Complete hematologic response (CHR)

    * No immature myeloid cells in peripheral blood
    * No increased basophils in peripheral blood
    * WBC less than upper limit of normal (ULN)
    * Platelet count less than ULN
    * No major (less than 35% Ph+) or complete (0% Ph+) cytogenetic response after at least 6 months of imatinib mesylate

      * Loss of prior major cytogenetic response or failure to achieve major cytogenetic response

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* See Disease Characteristics

Hepatic

* Bilirubin less than 1.5 times ULN
* AST or ALT less than 2.5 times ULN

Renal

* Creatinine less than 1.5 times ULN

Cardiovascular

* No New York Heart Association grade III or IV congestive heart failure
* No untreated symptomatic cardiac ischemia
* No underlying cardiac arrhythmia, including but not limited to any of the following:

  * Conduction abnormality/atrioventricular heart block
  * Nodal/junctional arrhythmia/dysrhythmia
  * Sinus bradycardia or tachycardia
  * Supraventricular tachycardia
  * Ventricular arrhythmia

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use 2 methods of effective barrier contraception during and for 3 months after study
* Electrolyte levels (especially potassium and magnesium) normal (CHR patients)
* No history of noncompliance that would preclude study participation
* No other concurrent serious, uncontrolled medical condition
* No grade 2 or greater neuropathy

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* More than 14 days since prior therapy except hydroxyurea, anagrelide hydrochloride, or imatinib mesylate
* More than 28 days since prior investigational agents
* No concurrent grapefruit or grapefruit juice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2002-10; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Satey and Tolerability
Dose-limiting toxicity
Pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: Michael Mauro, MD, Principal Investigator — OHSU Knight Cancer Institute
Locations (3):
- United States (3):
  - UCLA Department of Medicine, Division of Hematology/Oncology, Los Angeles, California
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - OHSU Knight Cancer Institute, Portland, Oregon